CLINICAL TRIAL: NCT01346891
Title: Polymorphisms of the Thiazide's Receptor Gene SLC12A3 and Development of Hyponatremia
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Sociedad Argentina de Hipertension Arterial (SAHA) (Other)
Responsible Party: Diego Giunta, Hospital Italiano de Buenos Aires
Other Study IDs: 1579
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-07

CONDITIONS: Thiazide Diuretics Induced Hyponatremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyponatremia Group (Cases): Patients over 21 years old, with confirmed antecedent of thiazide-induced hyponatremia who required hospitalization with a serum sodium concentration lower than 125 meq/L.
- Good Thiazide Tolerance (Controls): Patients over 21 years old, who have consumed thiazide diuretics for more than 2 years, with a serum sodium concentration persistently over 135 meq/L.

SUMMARY:
The purpose of this study is to detect if there are any differences in the coding region of SLC12A3 gene in individuals who have had hyponatremia associated to the use of thiazides, and those thiazides consumers without hyponatremia that have demonstrated good tolerance to the drug.

DETAILED DESCRIPTION:
This is a Case Control study to compare the coding region of SLC12A3 gene in individuals who have had hyponatremia associated to the use of thiazides, and those thiazides consumers without hyponatremia that have demonstrated good tolerance to the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 21 years, belonging to one of the following groups:

   1. Patients who have had Thiazide induced hyponatremia with serum sodium lower than 125 meq/L included in the Institutional Registry of Hyponatremia (Cases)
   2. Patients with good tolerance to chronic treatment with Thiazides tha never had associated hyponatremia (Controls)
2. Patients with normal serum sodium measurements before the start of the Thiazides

Exclusion Criteria:

1. Refusal to participate or to the informed consent process
2. Unclear cause of hyponatremia, or other hyponatremia cause concomitant to Thiazide diuretics
3. Patients related to other individuals already included in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 21 years old that require treatment with thiazide diuretics
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires F.D., Argentina